CLINICAL TRIAL: NCT04623996
Title: A Phase 1/2, Open-Label Clinical Study To Evaluate Safety And Efficacy Of TP-0184 To Treat Anemia When Administered To Adult Patients With IPSS-R Low Or Intermediate Risk Myelodysplastic Syndromes
Brief Title: A Study of TP-0184 to Treat Anemia in Adults With IPSS-R Low or Intermediate Risk MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to limitations imposed by the COVID pandemic and the competitive landscape for myelodysplastic syndrome, this study was unable to enroll a sufficient patient population.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI-TP-0184-102
Record Dates: First submitted 2020-10-20; First posted 2020-11-10 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Anemia in Myelodysplastic Syndromes
Keywords: Ph 1/2; Hematologic disease; MDS; Anemia; IPSS-R low; IPSS-R intermediate
MeSH Terms: conditions — Hematologic Diseases; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm TP-0184 (Experimental): TP-0184 is administered orally once a day
  Interventions: Drug: TP-0184

INTERVENTIONS:
Drug: TP-0184 — Oral dose

SUMMARY:
This study will evaluate preliminary safety and efficacy of TP-0184 to treat anemia when administered to adult patients with Revised International Prognostic Scoring System (IPSS-R) low or intermediate risk MDS. The recommended Phase 2 dose (RP2D) will be determined by the maximum tolerated dose (MTD) or maximum administered dose (MAD) in the Phase 1 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. A documented diagnosis of lower risk MDS (IPSS-R Low, Intermediate) according to WHO 2016 classification, de novo or secondary..
2. Bone marrow biopsy and/or aspirate performed pre-dose to assess disease status and available for review prior to full screening review. If the bone marrow biopsy and/or aspirate is nonproductive or nondiagnostic, the procedure must be repeated. Bone marrow biopsy/aspirate performed ≤ 12 weeks prior to baseline will not need to be repeated if results and a minimum of 6 slides are available.
3. Relapse, refractory/resistant, intolerant, or inadequate response to ESA treatment, as defined by the following:

   * Relapse according to IWG 2006
   * Refractory/resistant - documented non-response or response that is no longer maintained to prior ESA-containing regimen, either as single agent or combination (e.g., with G-CSF); ESA regimen must have been either:
   * Recombinant human erythropoietin (rHu EPO) ≥ 500 IU/wk for at least 8 doses or equivalent; OR
   * Darbepoetin alpha ≥ 300 μg Q3W for at least 4 doses or equivalent;
   * Intolerant- documented discontinuation of prior ESA containing regimen, either as single agent or combination (e.g., with G-CSF), at any time after introduction due to intolerance or an adverse event

   Inadequate response - in the absence of transfusions support, patients under ESA treatment for at least 12 weeks that do not show a rise in hemoglobin of greater than equal to 1 g/dl.
4. Patients with 5q deletions are allowed only if they have failed or are intolerant to lenalidomide treatment.

   o Failure or intolerance to lenalidomide defined as clinical and cytogenetic responses to according to the international working group 2006 MDS: (1) absence of response, or (2) bone marrow progression during treatment with or without prior response, or (3) secondary failure (loss of prior hematological response without bone marrow progression), or (4) intolerance (treatment discontinuation due to adverse events, with or without prior response) based on investigator judgement (Prebet 2017). 7
5. Patients previously treated for anemia with or without RBC transfusion support:

   1. Low transfusion burden (LTb), defined as requiring less than 4 red blood cell units in the 8 weeks before treatment (and baseline hemoglobin < 9.0 g/dL),
   2. High transfusion burden (HTb), defined as requiring 4 or more red blood cell units in the 8 weeks before treatment
6. At least 12 weeks of transfusion history immediately preceding the first dose of TP-0184. This transfusion data must include hemoglobin measured prior to transfusion (pre transfusion Hgb).
7. Written, signed consent for trial participation must be obtained from the patient appropriately in accordance with applicable ICH guidelines and local and regulatory requirements prior to the performance of any study specific procedure.
8. Must be ≥18 years of age.
9. Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score ≤ 2.
10. Patients with a life expectancy of ≥3 months (90 days) per the treating investigator.
11. Patients with adequate major organ functions meeting the following criteria on the basis of laboratory data within 28 days (4 weeks) before screening (if multiple data are available, most recent data during the period):

    1. Serum creatinine: ≤1.8 x the upper limit of the normal (ULN) range
    2. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except in patients with Gilbert's syndrome. Patients with Gilbert's syndrome may enroll if direct bilirubin ≤2.0 x ULN or if the elevated total bilirubin can be attributed to active red blood cell precursor destruction within the bone marrow (i.e., ineffective erythropoiesis). Elevated indirect bilirubin due to post-transfusion hemolysis is allowed.
    3. Aspartate transaminase (AST) and alanine transaminase (ALT): ≤2.5 x ULN

    Left ventricular ejection fraction (LVEF) ≥ 45% by echocardiogram or multigated acquisition (MUGA) scan
12. All previous therapy with ESAs, G-CSF and GM-CSF must be discontinued ≥ 14 days before Cycle 1 Day 1 dosing.
13. Twenty-eight-day (4 weeks) washout period from prior treatment with cytotoxic chemotherapeutic agents, HMAs (hypomethylating agents), ImiDs (immunomodulatory imide drugs), luspatercept and / or investigational drugs before study dosing for the patient begins.
14. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 5 days prior to the first dose of TP-0184.
15. Non-fertile or agree to use an adequate method of contraception while on study and for 7 months following the study and have a negative pregnancy test (if female of childbearing potential) and not currently nursing; males agree to use an adequate method of contraception while on study and for 4 months following the study.
16. Patients must be able to comply with the requirements of the entire study and accessible for treatment and follow-up.
17. Patient agrees not to participate in other interventional clinical studies during their participation in this trial, while on study treatment. Patients participating in surveys or observational studies are eligible to participate in this study.

Exclusion Criteria:

1. IPSS-R high or very high risk MDS.
2. Presence of concomitant severe cardiovascular disease; congestive heart failure (CHF), myocardial infarction, angina and/ or uncontrolled cardiac arrhythmia as determined by the investigator within 6 months (180 days) of study onset.
3. Corrected QT interval (using Fridericia's correction formula) of > 465 msec in men and > 480 msec in women.
4. History of stroke, deep venous thrombosis (DVT), pulmonary or arterial embolism within 6 months (180 days) prior to enrollment.
5. Presence of clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding.

   a. Iron deficiency to be determined by a bone marrow aspirate stain for iron, calculated transferrin saturation (iron/total iron binding capacity) ≤ 20%, or serum ferritin ≤ 15 µg/L.

   b. Iron-chelating agents, except for subjects on a stable or decreasing dose for at least 8 weeks prior to enrollment, are excluded
6. Prior allogeneic or autologous stem cell transplant due to myeloid disease
7. Known history of diagnosis of AML.
8. Use of corticosteroid, except for subjects on a stable or decreasing (no greater than a 10 mg dose of prednisone or equivalent) for ≥ 2 weeks prior to enrollment for medical conditions other than MDS
9. Patients are excluded if there is evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count (reticulocyte index) of > 2% with either a positive Coombs' test or over 50% indirect bilirubin.
10. Patients with a recent diagnosis of malignancy are excluded except for those with in situ malignancies treated with curative intent (eg, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix). Patients with more advanced malignancies are allowed to enroll, provided they were treated with curative intent and have no evidence of active disease ≥ 2 years prior to Cycle 1 Day 1.
11. Patients requiring systemic antibiotics or antifungals are not eligible until they have completed the prescribed course of antibiotics or antifungals and are clinically stable. Topical antibiotics or antifungals are permitted.
12. Known HIV, active Hepatitis B, and/or active Hepatitis C infection.
13. Patients with clinically active uncontrolled, bleeding in the past month.
14. Thrombocytopenia (platelet count < 50,000/µL [50 x 109/L]).
15. Neutropenia (absolute neutrophil count [ANC] <500 /µL [0.5 x 109/L])
16. Women who are pregnant or breastfeeding.
17. Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second effective method of contraception during the trial and for 7 months after the last administration of study treatment.
18. Inability to undergo MRI imaging.
19. Parenchymal iron overload by screening MRI.
20. Patients who are unwilling or unable to comply with procedures required in this protocol.
21. Have undergone recent surgery with potential to cause the impairment of gastrointestinal tract absorption or that could cause short bowel syndrome with diarrhea due to malabsorption.
22. Have known hemochromatosis at baseline or a family history of hemochromatosis.
23. Presence of any psychological, familial, sociological or geographical condition that, in the opinion of the investigator, could potentially hinder compliance with the study protocol and follow-up schedule.
24. Patient has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
25. Live vaccines within 14 days prior to first study drug administration. COVID-19 vaccines (non-live) approved by regional health authorities are allowed.
26. Medications that are known strong to moderate CYP3A4 inducers must be discontinued at least 21 days prior to first dose of study drug. Medications that are known strong to moderate CYP3A4 inhibitors must be stopped 21 days (or 5 half-lives, whichever is shorter) prior to the first dose of study drug.
27. Patients who have received medications with known or possible risk of prolonging the QT interval or inducing Torsades de Pointes within the previous 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - BRCR Global, Plantation, Florida
  - Montefiore Medical Center, The Bronx, New York
  - US Oncology - Austin Texas Oncology Midtown, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to limitations imposed by the COVID pandemic and the competitive landscape for myelodysplastic syndrome, this study was unable to enroll a sufficient patient population. The decision was made to terminate the study early and discontinue further development of the TP-0184 program. The 2 patients enrolled into phase 1 of the study withdrew their consent to participate on 30 March 2021 and 27 April 2021; no further patients were enrolled.
Pre-assignment Details: Participants who died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Phase 1: Single Arm TP-0184: Participants who were enrolled to phase 1 received TP-0184, with starting dose of 20mg, administered orally, once daily, following an overnight fast of at least 6 hours.
- Phase 2: Single Arm TP-0184: Participants who were enrolled to phase 2 would receive the recommended phase 2 dose (RP2D) as determined in phase 1.
Period: Overall Study
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The company decided to terminate further development of the TP-0184 program. No patients were enrolled into phase 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184 | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Full Range); unit: years] | 63 [44 to 82] |  | 63 [44 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Tolerability of TP-0184 as Evaluated by Incidence of Dose Limiting Toxicities (DLTs) as Observed in Cycle 1
Description: DLTs are defined as follows: Any Gr 3 or greater nonhematologic toxicity; New onset cardiac failure or worsening symptomatic cardiac failure; Echocardiogram (ECHO) or multigated acquisition (MUGA) reduction of ejection fraction (EF) > 10%; Any Gr 4 neutropenia; Any Gr 3 thrombocytopenia associated with clinically significant bleeding, or Gr 4 thrombocytopenia in the absence of myelodysplasia-related marrow failure or transformation to acute leukemia; All other hematologic toxicity Grade 3 or higher other than defined above for ANC or platelets
Time Frame: Cycle 1 (28 days)
Population: Sponsor's decision to terminate further development of the TP-0184 program. Data collection and analysis were therefore not conducted as planned.
Arm/Group | Phase 1: Single Arm TP-0184
Number analyzed (Participants) | 0

2. Primary Outcome: Phase 1: Number of Participants With Adverse Events and Serious Adverse Events
Description: Assessment of safety of TP-0184 administered in participants by reporting of adverse events and serious adverse events
Time Frame: The time from the date of first treatment, while the patient is taking TP-0184, and for 30 days after stopping therapy, an average of 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Single Arm TP-0184
Number analyzed (Participants) | 2
Participants | 2

3. Primary Outcome: Phase 2: The Effect of TP-0184 on the Treatment and the Hematologic Improvement of Anemia in Terms of Hemoglobin Increase, Reduction in RBC Transfusions and Transfusion-free Equal or Greater Than 8 Weeks
Description: Response rate based on composite response criteria: Hemoglobin increase greater than or equal to 1.5 g/dL, maintained for a consecutive period of 8 weeks with no transfusions; OR reduction in units of greater than or equal to 4 RBC transfusions / 8 weeks (consecutive) compared with the pretreatment transfusion number in previous 8 weeks; OR patients who are RBC transfusion-free over any consecutive 8-week (56-day) period
Time Frame: 56 days
Population: Sponsor's decision to terminate further development of the TP-0184 program. Data collection and analysis were therefore not conducted as planned. No patients were enrolled into phase 2.
Arm/Group | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1: The Effect of TP-0184 on the Treatment and the Hematologic Improvement of Anemia in Terms of Hemoglobin Increase, Reduction in RBC Transfusions and Transfusion-free Equal or Greater Than 8 Weeks
Description: as for outcome 3
Time Frame: 56 days
Population: as for outcome 1
Arm/Group | Phase 1: Single Arm TP-0184
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 1/2: The Effect of TP-0184 on the Treatment and the Hematologic Improvement of Anemia in Terms of Hemoglobin Increase, Reduction in RBC Transfusions and Transfusion-free Equal or Greater Than 12 Weeks
Description: Response rate based on composite response criteria: Hemoglobin increase greater than or equal to 1.5 g/dL, maintained for a consecutive period of 12 weeks with no transfusions; OR reduction in units of greater than or equal to 4 RBC transfusions / 12 weeks (consecutive) compared with the pretreatment transfusion number in previous 12 weeks; OR patients who are RBC transfusion-free over any consecutive 12-week (84-day) period
Time Frame: 84 days
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 1/2: Determine the Time to RBC Transfusion-free Period
Description: Time from first dose of TP-0184 to the first onset of a transfusion-free period for consecutive 8 weeks
Time Frame: 56 days
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 1/2: Determine the Median Duration of Hemoglobin Response
Description: Duration of hemoglobin increase greater or equal to 1.5 g/dL maintained for a consecutive period of > 8 weeks with no transfusions.
Time Frame: 56 days
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase 1/2: Determine the Median Duration of Reduction in RBC Transfusions
Description: Duration of reduction in units of greater or equal to 4 RBC transfusions / 8 weeks (consecutive)
Time Frame: 56 days
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase 1/2: Determine the Median Duration of RBC-transfusion-free Period Greater or Equal to 8 Weeks
Description: Duration of RBC transfusion-free period
Time Frame: 56 days
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 1/2: Determine the Cardiac Safety of TP-0184 by Assessing the Presence of Cardiac Symptoms
Description: Assessment of cardiac safety of TP-0184 administered in participants by reporting of cardiac symptoms including congestive heart failure (CHF). Assessment of CHF will be based based on NYHA criteria, 12-Lead ECG abnormalities, quantification of cardiac iron by MRI, ECHO or MUGA scans, and peripheral blood cardiac markers
Time Frame: as for outcome 2
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Phase 1/2: Determine the Proportion of Patients Progressing to AML
Description: Proportion of patients progressing to AML
Time Frame: 4 months
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase 1/2: Determine Overall Survival
Description: The effect of TP-0184 on the overall survival
Time Frame: From the first dose of TP-0184 until the time of death due to any cause, up to 4 months off treatment.
Population: as for outcome 3
Arm/Group | Phase 1: Single Arm TP-0184 | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Phase 1: Determination of the Maximum Observed Concentration (Cmax) and Area Under the Plasma Concentration vs. Time Curve (AUClast)
Description: To determine the maximum concentration of TP-0184 and the area under the plasma concentration vs. time curve of TP-0184
Time Frame: Phase 1: Blood samples drawn on days 1, 2, 4, 8, 15, and 22 of the first study cycle; days 1, 8, 15, and 16 of the 2nd cycle. Phase 2: Blood samples drawn on Cycle 1, day 22; cycle 2, days 1, 8 and 15; cycle 3, day 1.
Population: as for outcome 1
Arm/Group | Phase 1: Single Arm TP-0184
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 2: Determine the Changes in Neutrophil Counts
Description: Proportion of patients achieving hematologic improvement in neutrophil count (HI-N) over any consecutive 8-week (56-day) period and / or decrease in neutrophil count
Time Frame: 56 days
Population: Sponsor's decision to terminate further development of the TP-0184 program. Data collection and analysis were therefore not conducted as planned. No patients enrolled into phase 2.
Arm/Group | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 2: Determine the Changes in Platelet Counts
Description: Proportion of patients achieving hematologic improvement in platelets (HI-P) over any consecutive 8-week (56-day) period and / or decrease in platelet count
Time Frame: 56 days
Population: as for outcome 3
Arm/Group | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 2: Number of Participants With Adverse Events (AEs) & Serious Adverse Events (SAEs)
Description: Assessment of safety and tolerability of TP-0184 administered in participants by reporting of AEs and SAEs
Time Frame: The time from the date of first treatment, while the patient is taking TP-0184, and for 30 days after stopping therapy, up to 6 months.
Population: as for outcome 14
Arm/Group | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 2: Determine Steady-state Trough PK
Description: Characterize TP-0184 plasma trough concentration data at various timepoints.
Time Frame: Cycle 1 Day 1 of Week 4 and Cycle 2 Day 1 of each Week 5, 6, 7, and 9
Population: as for outcome 3
Arm/Group | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0

18. Secondary Outcome: Phase 2: Determine the Level of Fatigue Based Off of the Brief Fatigue Inventory (BFI)
Description: The BFI measures the severity of fatigue based on the worst fatigue experienced during the past 24-hours
Time Frame: From the first dose of TP-0184 up to 4 months or study closure
Population: as for outcome 3
Arm/Group | Phase 2: Single Arm TP-0184
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death or withdrawal of consent, up to 4 months off treatment.
Description: Sponsor's decision to terminate further development of the TP-0184 program. No patients were enrolled into phase 2.
Arm/Group | Phase 1: Single Arm TP-0184
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Single Arm TP-0184 (N=2)
overdose (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Single Arm TP-0184 (N=2)
nausea (Gastrointestinal disorders) | 1
diarrhoea (Gastrointestinal disorders) | 1
fatigue (General disorders) | 2
headache (Nervous system disorders) | 1
vision blurred (Eye disorders) | 1
abdominal pain (Gastrointestinal disorders) | 1
dyspepsia (Gastrointestinal disorders) | 1
ageusia (Nervous system disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 2
anosmia (Nervous system disorders) | 1
chills (General disorders) | 1
decreased appetite (Metabolism and nutrition disorders) | 1
SARS-CoV-2 test positive (Investigations) | 2
dry eye (Eye disorders) | 1
dysuria (Renal and urinary disorders) | 1
Klebsiella infection (Infections and infestations) | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 1
pollakiuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT04623996/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT04623996/SAP_001.pdf